CLINICAL TRIAL: NCT05743283
Title: Efficacy of SynEx™ Wound Rinse in Civilian Surrogates of Combat Injury Wounds
Brief Title: Efficacy of SynEx Wound Rinse in Civilian Surrogates of Combat Injury Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Synedgen, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency); Medical Technology Enterprise Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SynEx
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Wound Heal
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel-group, comparator-controlled interventional study to assess clinical efficacy of SynEx Wound Cleanser.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SynEx (Experimental): The experimental arm will receive SynEx Wound Cleanser to cleanse the wound as directed by their healthcare provider.
  Interventions: Device: SynEx Wound Cleanser
- Saline (Active Comparator): The comparator arm will receive Saline Solution to cleanse the wound as directed by their healthcare provider.
  Interventions: Other: Saline

INTERVENTIONS:
Device: SynEx Wound Cleanser — SynEx is a concentrated form of SynePure®, an FDA 510(k) cleared aqueous, osmotically balanced wound cleanser containing patented chitosan derivatives. The ingredients are USP purified water, chitosan arginine (a patented chitosan derivative), sorbitol powder, and betaine. SynEx cleanser is packaged in a collapsible plastic pouch for reconstitution in water before debriding and cleansing a wound.
  Arms: SynEx
Other: Saline — The saline solution is composed of water and salt. It is packaged in a collapsible plastic pouch.
  Arms: Saline

SUMMARY:
The purpose of this interventional study is to compare SynEx Wound Cleanser with the current routine care (Saline) in traumatic wounds. Participants with gunshot, penetrating or burn wounds who participate will be asked to attend up to four study visits, use the assigned wound cleanser and complete brief surveys about their healing and well-being related to the wound healing.

ELIGIBILITY:
Inclusion Criteria:

1. Acute penetrating, puncture and burn wounds of the upper or lower extremity that meet the inclusion and exclusion criteria for the wound type:

   1. Penetrating, puncture or laceration wounds: stage II-III (partial to full thickness loss of dermis) excluding diabetic or venous wounds, and pressure ulcers and perforated wounds (except gunshot wounds) and wounds with exposed bones, facia or muscle.
   2. Gunshot wounds (GSW): Grade I - II on the Red Cross Classification of War Wounds6 (diameter of entry + exit wounds < 10 cm, wound cavity or not, no fracture or fraction without clinically significant comminution). Non-penetrating, penetrating, or perforated GSW are included. GSW with suspected vascular injuries or nerve damage are excluded.
   3. Burns: partial thickness injury ≤ 9% TBSA. Thermal burn from flame or scald, chemical burns, and electrical burn are included. Radiation and frostbite burns are excluded.
2. Males and females ≥18 years old.
3. Has access to a computer or mobile device for telepresence visits.
4. Able to give informed consent and willing to comply with all required study procedures.

Exclusion Criteria:

1. Any wound likely to require irrigation and debridement in an operating room (OR) setting.
2. Concomitant processes sustained contemporaneously with the dermal injury (e.g., inhalational injury requiring ventilation, electrical injury with cardiac damage or arrhythmia, sepsis, traumatic brain injury, other serious or unstabilized organ damage from trauma, etc.).
3. > 72 hrs from initial injury.
4. Pregnant or lactating females.
5. Patients with known allergy(ies) to any of the components of the study irrigation system.
6. Patients who are considered by the investigator for any reason to be an unsuitable candidate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Wound healing environment composite score | 14 days
  The composite score is a summation of wound characteristics such size, depth, edges and undermining. Scores range from range of 13 to 60, representing wound regeneration to degeneration respectively).

CONTACTS AND LOCATIONS:
Overall Officials: Shenda Baker, PhD, Principal Investigator — Synedgen, Inc.
Locations (2):
- United States (2):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Barnes Jewish Hospital, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No